CLINICAL TRIAL: NCT03649789
Title: Retrospective Study of Periodontal Outcomes After Sanative Therapy in Patients With or Without Salivary Gland Hypofunction
Brief Title: Periodontal Outcomes After Sanative Therapy
Status: Completed | Type: Observational
Sponsor: Brock University (Other)
Collaborators: Dr. Peter C. Fritz, Periodontal Wellness & Implant Surgery (Other)
Responsible Party: Principal Investigator, Wendy E. Ward, Ph.D., Professor and Canada Research Chair, Brock University
Other Study IDs: 17-387-WARD
Record Dates: First submitted 2018-07-19; First posted 2018-08-28 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Periodontal Pocket; Xerostomia; Dry Mouth; Periodontal Diseases
Keywords: healing; biomarkers; sanative therapy; nutritional supplements; medications; salivary flow
MeSH Terms: conditions — Periodontal Pocket; Xerostomia; Periodontal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Saliva is being collected at time of hygiene appointment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No Salivary Gland Hypofunction: These individuals have an unstimulated salivary flow rate of greater than 0.1 mL saliva/min.
- Salivary Gland Hypofunction: These individuals have an unstimulated salivary flow rate of less than 0.1 mL saliva/min.

SUMMARY:
Salivary gland hypofunction, or dry mouth, is a damaging oral condition that affects salivary gland production. Absence of saliva causes bad breath, dental decay, increased plaque accumulation, dry lips, mouth sores, and the inability to retain dentures or removable protheses. This study will determine if patients with dry mouth have different periodontal health than patients without dry mouth. Additionally, this study will examine if patients who have their periodontal maintenance appointments solely at a periodontal speciality clinic have different periodontal health than patients who alternate their appointments between a specialty office and their general dental office.

DETAILED DESCRIPTION:
Salivary gland hypofunction, or dry mouth, is a damaging oral condition that affects the function and flow rate of saliva. Low saliva rates can range from mild self-reported symptoms and discomfort to significant oral diseases. Saliva is essential in preventing irritation and friction of mucosal surfaces. Progressively dry mouth can cause oral and bodily conditions that can affect an individuals quality of life and daily tasks, such as eating and avoiding social situations. Specifically, dry mouth is a risk factor for periodontal disease, a chronic oral inflammation of tissues and ligaments that support the tooth's structure and if untreated, will ultimately lead to tooth loss. In Canada, the first line of defense against periodontal disease is non-surgical sanative therapy (ST). Participants in this study have been attending a periodontal specialty clinic for routine periodontal maintenance appointments for at least 1 to 5 years following their initial scaling and root planing. Salivary flow rate will be measured to determine the level of dry mouth. At the regular maintenance appointment, clinical measures will be evaluated (probing depth, bleeding on probing, plaque index, gingival index, thickness of tissues, mobility, and furcations). Patients will also complete a dry mouth questionnaire to determine if dry mouth influences the day to day life of a patient, and the patient's Registered Dental Hygienist will complete a short questionnaire outlining oral symptoms of dry mouth. Additionally, the investigators aim to see if a patient who has periodontal maintenance appointments at a specialty office has different clinical outcomes than a patient who alternates these appointments between a specialty office and a general dental office. Overall, the investigators will determine if thorough periodontal maintenance appointments are efficient in preventing periodontal disease in patients with dry mouth.

ELIGIBILITY:
Inclusion Criteria:

* have had sanative therapy at this clinic in the previous 1 to 5 years.

Exclusion Criteria:

* anyone who is unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who previously underwent sanative therapy to manage periodontal disease at this clinic and who have regular maintenance periodontal cleanings on a regular basis at the clinic.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Probing Depth | At maintenance appointment (1 hour) and retrospectively from the clinical record from time of sanative therapy onwards
  Probing depth is a routine clinical measure of periodontal health (measured in mm)

SECONDARY OUTCOMES:
Bleeding on Probing | At maintenance appointment (1 hour) and retrospectively from the clinical record from time of sanative therapy onwards
  Bleeding on Probing is a measure of inflammation and determined as the percent of bleeding sites that are measured at 6 sites per tooth.
O'Leary Index of Plaque Control | At maintenance appointment (1 hour) and retrospectively from the clinical record from time of sanative therapy onwards
  The patient's plaque index = the number of plaque-containing surfaces divided by the total number of available surfaces.
  For instance, if a patient has 28 teeth they have 112 tooth surfaces (28x4=112) and if 40 surfaces contain plaque their plaque index is 40/112=0.357 or 35.7%.
  The minimum plaque index would be 0%, which represents no tooth surfaces that contain plaque.
  The maximum plaque index would be 100%, which represents all surfaces of the patient's teeth contain plaque.
  The optimal outcome is to have a plaque index of 0%. The worst outcome would be a plaque index of 100%.
Gingival Index (used to assess gingival condition to distinguish between the quality of gingiva and the location of gingival concerns). | At maintenance appointment (1 hour) and retrospectively from the clinical record from time of sanative therapy onwards
  The gingival index system consists of 4 possible ratings: 0 = Normal gingiva, 1 = mild inflammation with a slight change in colour, slight edema (no bleeding on probing); 2 = moderate inflammation with redness, edmea and glazing (bleeding on probing); or 3 = severe inflammation with marked redness and edema, ulceration, tendency to spontaneous bleeding.
  Each four gingival areas of a tooth is given a score from 0 to 3. This corresponds to the gingival index for that area.
  The scores from the four areas of the tooth can be added and divided by four to give the gingival index for the tooth.
  The better outcome is having a gingival index of 0, the worst outcome is having a gingival outcome of 3.
Thickness of Periodontal Tissue | At maintenance appointment (1 hour)
  Assessment of gingival tissue thickness to assess tissue quality and response to inflammation
Body Mass Index (BMI) | At maintenance appointment (1 hour)
  Assessment of body weight and height to calculate BMI as it is a known risk factor for periodontal disease
Dry Mouth Inventory Questionnaire Completed by the Patient (to assess impact of dry mouth on quality of life) | At maintenance appointment (1 hour)
  This questionnaire measures, at one time point, the self-reported daily limitations due to dry mouth. This inventory questionnaire includes 11 criteria and the questionnaire is completed by the patient.
  The 11 criteria include: I sip liquids to aid in swallowing food; My mouth feels dry when eating a meal; I get up at night to drink; My mouth feels dry; I have difficulty in eating dry foods; I suck sweets or cough lollies to relieve dry mouth; I have difficulties swallowing certain foods; The skin on my face feels dry; My eyes feel dry; My lips feel dry; The inside of my nose feels dry.
  For each of the criteria, patients will also rate the frequency by which having a dry mouth limits their daily functions according to the following description: "never", "hardly ever", "occasionally", "fairly often", "very often"
The Hygienist Observational Symptom Questionnaire (to assess whether a patient has dry mouth) | At maintenance appointment (1 hour)
  The hygienist records the following about their patient using this questionnaire:
  * Symptoms of dry mouth identified using the following criteria: patient's initial salivation volume and consistency as copious, adequate, slight, or deficient in volume as well as if the consistency is serous, sticky, or frothy. Best outcome is a copious salivary volume and a saliva consistency that is serous. Worst outcome is a deficient saliva volume and a consistency of saliva that is frothy.
  * Record presence of dental caries, enamel demineralization, tooth hypersensitivity, mucositis, oral candidiasis, traumatic gingival ulcerations, fissure tongue, crenulations on tongue, dry lips, angular chelitis, halitosis, food retention on teeth and/or tongue, or loss of papilla on tongue. All listed outcomes would be considered worst outcomes of dry mouth. Patients would benefit from having none of the above.
  * Record use of any current treatment for dry mouth.
Frequency of Periodontal Maintenance Appointment at the Periodontal Clinic and General Dental Clinic | Will be reviewed from patient's clinical record over a time period of 1 to 5 years (this will represent the time period from recruitment and retrospectively until the time at which sanative therapy was performed)
  Frequency of periodontal maintenance appointments at the periodontal clinic and general practice will be recorded.
Frequency of Periodontal Maintenance Appointment only at the Periodontal Clinic | Will be reviewed from patient's clinical record over a time period of 1 to 5 years (this will represent the time period from recruitment and retrospectively until the time at which sanative therapy was performed)
  Frequency of periodontal maintenance appointments at the periodontal clinic will be recorded.

OTHER OUTCOMES:
Furcations | At maintenance appointment (1 hour) and retrospectively from the clinical record from time of sanative therapy onwards
  Furcations are classified (Class 1 through 3) as amount of bone loss surrounding the root of a tooth.
Tooth Mobility | At maintenance appointment (1 hour) and retrospectively from the clinical record from time of sanative therapy onwards
  Tooth Mobility is classified (Class 1 through 3) as amount of support around a tooth.
Salivary Markers of Inflammation | At maintenance appointment (1 hour)
  Specific markers of inflammation measured in saliva
Dietary Supplement Intakes | At maintenance appointment (1 hour) and retrospectively from the clinical record from time of sanative therapy onwards
  Intakes of specific dietary supplements measured using a dietary supplement questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Wendy E Ward, PhD, Principal Investigator — Brock University
Locations (2):
- Canada (2):
  - Dr. Peter C. Fritz, Periodontal Wellness & Implant Surgery, Fonthill, Ontario
  - Brock University, St. Catharines, Ontario

IPD SHARING:
Plan to Share IPD: Undecided